CLINICAL TRIAL: NCT07205731
Title: PRODIGE 102 - FFCD 2201 - SAFE-ESO Phase II Study Evaluating Safety and Efficacy of Tislelizumab for Elderly Patients Unfit for Chemotherapy, With Advanced Esophageal Squamous-cell Carcinoma
Brief Title: Phase II Study Evaluating Safety and Efficacy of Tislelizumab for Elderly Patients Unfit for Chemotherapy, With Advanced Esophageal Squamous-cell Carcinoma
Acronym: SAFE ESO
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: BeiGene USA, Inc. (Industry); Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PHRC K 2023 JARY
Record Dates: First submitted 2025-09-12; First posted 2025-10-03 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2026-01

CONDITIONS: Esophageal Squamous Cell Carcinoma (ESCC)
Keywords: digestive oncology; immunotherapy; microenvironment biomarker; oncology; oncogeriatric domain; Ederly patients; chemotherapy
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- all patients receive the Tislelizumab on monotherapy (Experimental)
  Interventions: Drug: Tislelizumab is a fully humanized monoclonal antibody specific for human PD-1

INTERVENTIONS:
Drug: Tislelizumab is a fully humanized monoclonal antibody specific for human PD-1 — It is the first study which evaluate efficacy and safety of anti PD-1 immune checkpoint inhibitor alone in the first-line treatment of elderly esophageal squamous-cell carcinoma patients who no fit to received chemotherapy with platine

SUMMARY:
The goal of this clinical trial is to assess the percentage of patients alive at 6 months in elderly patients, not eligible to an platinum-based chemotherapy, but who can received the Tislelizumab treatment alone as first-line treatment for an advanced esophageal squamous-cell carcinoma (ESCC).

Tislelizumab is a monoclonal antibody administred by intravenous infusion

This study aims to anwer too at the questions:

* the Safety of the drug
* Overall survival (OS) at 6 months according the diagnostic of PD-L1 expression (PD-L1 is a protein present on the surface of immune cells)
* Overall response rate (ORR) according to imagery criteria
* Progression-free survival (PFS) at 3 and 6 months according to imagery criteria and depending on PDL1 expression
* Patients' health-related quality of life
* OS and PFS according to geriatric parameters
* Prognostic value of immune biomarkers

DETAILED DESCRIPTION:
This is a multicenter open-label single arm phase II study to evaluate Tislelizumab in monotherapy in frontline metastatic or locally advanced ESCC.

Patient aged ≥70 years will be selected for inclusion after a diagnosis of metastatic or locally advanced ESCC, and if they are not eligible for a platinum-based chemotherapy regimen.

Tislelizumab (200 mg flat dose every 3 weeks) will be received by intravenous perfusion until progression or unacceptable toxicity, for a maximum of 2 years.

The patients will be included regardless of PD-L1 status; A comparison for all study population will be carried out centrally as part of the ancillary enquiries.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven esophageal squamous cell carcinoma (ESCC)
* Metastatic or locally advanced cancer
* Absence of previous treatment (immunotherapy, chemotherapy or radiotherapy) in first line setting
* Ineligibility for a platinum-based chemotherapy assessed by oncologist and geriatrician
* At least one evaluable and/or measurable lesion as defined by RECIST v1.1 criteria
* Patients ≥ 70 years
* Subjects with WHO performance status ≤ 2
* Estimated life expectancy >3 months
* Adjuvant therapy finished >6 months
* Adequate marrow and organ functions defined as:

  * Absolute neutrophil count (ANC) ≥ 1 × 109/L,
  * Platelet count ≥ 75 × 109/L,
  * Hemoglobin ≥ 90 g/L,
  * Aspartate transaminase (AST) and alanine transaminase (ALT) ≤ 3 × ULN, or AST and ALT ≤5 ×ULN for patients with liver metastases
  * ALP ≤ 5 x ULN unless liver metastases are present, in which case it must be ≤ 10x ULN
  * Measured creatinine clearance (CL) > 40 mL/min (MDRD method)
* Male patients must use a condom during treatment and for 6 months after the last dose when having sexual intercourse with a pregnant woman or with a woman of childbearing potential. Female partners of male patients should also use a highly effective form of contraception if they are of childbearing potential during treatment and for 6 months after the last dose.
* Patient is willing and able to comply with the protocol for the duration of the study including undergoing treatment, scheduled visits and examinations including follow up.
* Signed written informed consent obtained prior to any study specific procedures
* Patient affiliated to a social security scheme

Exclusion Criteria:

* History of another primary malignancy. May be included, patients with:

  * Malignancy treated with curative intent and with no known active disease ≥ 2 years before the first dose of treatment
  * Adequately treated non-melanoma skin cancer or lentigo maligna without evidence of disease
  * Adequately treated carcinoma in situ without evidence of disease
* Locally advanced esophageal carcinoma that is resectable or potentially curable with radiation therapy per local investigator
* Participation in another clinical study with an investigational product during the last 2 months.
* Concurrent enrolment in another clinical study unless it is an observational (non-interventional) clinical study or during the follow-up period of an interventional study.
* History of allogenic organ, bone marrow, or double umbilical cord blood transplantation
* Active documented autoimmune or inflammatory disorders (including inflammatory bowel disease [e.g., colitis or Crohn's disease], systemic lupus erythematosus, Sarcoidosis syndrome, or Wegener syndrome [granulomatosis with polyangiitis, Graves' disease, rheumatoid arthritis, hypophysitis, uveitis, etc]). May be included:

  * Patients with vitiligo or alopecia
  * Patients with hypothyroidism (e.g., following Hashimoto syndrome) stable on hormone replacement.
  * Any chronic skin condition that does not require systemic therapy.
  * Patients with celiac disease controlled by diet alone
* Previous immune checkpoint inhibitor therapy within the 2 years before inclusion
* Uncontrolled intercurrent illness; uncontrollable pleural effusion, pericardial effusion, or ascites requiring frequent drainage or medical intervention (recurrence ≤ 14 days after intervention). Patients with the following diseases are not excluded and may proceed to further screening:

  * Controlled Type I diabetes
  * Hypothyroidism (provided it is managed with hormone replacement therapy only)
  * Controlled celiac disease
  * Skin diseases not requiring systemic treatment (eg, vitiligo, psoriasis, alopecia)
  * Any other disease that is not expected to recur in the absence of external triggering factors
* Patients with evidence of fistula (either oesophageal/bronchial or oesophageal/aorta)
* Patients considered at poor medical risk due to a serious, uncontrolled medical disorder, non-malignant systemic disease, or active, uncontrolled ventricular arrhythmia, recent (within 6 months) myocardial infarction, pulmonary embolism/deep vein thrombosis, cerebrovascular accident, and heart failure, uncontrolled major seizure disorder, unstable spinal cord compression, superior vena cava syndrome, interstitial bilateral lung disease on high Resolution Computed Tomography (HRCT) scan or any psychiatric disorder that prohibits obtaining informed consent. Underlying medical conditions (including laboratory abnormalities) or alcohol or drug abuse or dependence that will be unfavorable for the administration of study drug or affect the explanation of drug toxicity or AEs or might impair compliance with study conduct. A history of severe hypersensitivity reactions to other monoclonal antibodies. Has received any chemotherapy, immunotherapy (eg, interleukin, interferon, thymosin, etc) or any investigational therapies within 14 days or 5 half-lives (whichever is shorter) of the first study drug administration.
* Patients with myelodysplastic syndrome/acute myeloid leukaemia or with features suggestive of MDS/AML.
* Patient with symptomatic central nervous system (CNS) metastases.
* History of active primary immunodeficiency.
* Known non-controlled serologically positive human immunodeficiency virus (HIV) patients with CD4 < 400 / mm3.
* Active infection including tuberculosis (clinical evaluation that includes clinical history, physical examination and radiographic findings, and TB testing in line with local practice), active untreated hepatitis B (known positive HBV surface antigen (HBsAg) result), active untreated hepatitis C. Patients with a past or resolved HBV infection (defined as the presence of hepatitis B core antibody [anti-HBc] and absence of HBsAg) are eligible. Patients positive for hepatitis C (HCV) antibody are eligible only if polymerase chain reaction is negative for HCV RNA.
* Current or prior use of immunosuppressive medication within 14 days before the first dose of -immunotherapy. The following are exceptions to this criterion:

  * Intranasal, inhaled, topical steroids, or local steroid injections (e.g., intra articular injection)
  * Systemic corticosteroids at physiologic doses not to exceed 10 mg/day of prednisone or its equivalent
  * Steroids as premedication for hypersensitivity reactions (e.g., CT scan premedication)
* Receipt of live attenuated vaccine within 30 days prior to the first dose of ICI
* Follow-up impossible, according to investigator's decision
* Any psychological, familial, sociological, or geographical condition potentially hampering compliance with the study protocol or follow-up schedule
* Persons i) deprived of liberty by judicial or administrative decision, persons subject to psychiatric care under Articles L. 3212-1 and L. 3213-1 who do not fall under the provisions of Article L. 1121-8 and persons admitted to a health or social care facility for purposes other than research, and (ii) adults subject to a legal protection measure or unable to express their consent (Article L1121-8)

Min Age: 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 95 (Estimated)
Dates: Start 2025-10-07 (Actual); Primary Completion 2029-10 (Estimated); Study Completion 2030-10 (Estimated)

PRIMARY OUTCOMES:
To assess the percentage of patients alive at 6 months in elderly patients, not eligible to platinum-based chemotherapy, treated by anti-PD1 Tislelizumab alone as first-line treatment for an advanced ESCC | 6 month after inclusion
  to assess the rate of evaluable patients (i.e., those not lost to follow-up at 6 months and who have received at least one dose of the study treatment) who are alive at 6 months after inclusion to patient rate measurement

SECONDARY OUTCOMES:
Safety according to NCI-CTCAE version 5.0 | time between the date of the first dose treatment with tislelizumab and the date within the 90 days after the last dose of treatment
  all grade and severe (grade 3-5) toxicities, according to the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0, will be recorded until 90 days after the last administration of treatment
- Overall survival (OS) at 6 months depending on PD-L1 expression | time between the date of the first dose treatment with tislelizumab and the date of death (whatever the cause) or date of last news for alive patients
  Overall survival (OS) will be estimated by the time between the date of the first dose treatment with tislelizumab and the date of death (whatever the cause) or date of last news for alive patients
- Overall response rate (ORR) according to RECIST 1.1 criteria | the time between the date of the first dose treatment with tislelizumab and the date of last dose of treatment
  The Overall Response Rate (ORR): is defined as the proportion of patients who achieved complete response (CR) or partial response (PR) as the best response during the treatment. evaluated by the investigator according to RECIST 1.1 criteria.
Progression-free survival (PFS) at 3 and 6 months according to RECIST 1.1 criteria and depending on PDL1 expression | at 3 month and 6 month after inclusion
  Progression free survival (PFS) is defined by the time between the date of the first dose treatment with tislelizumab and the date of first progression (clinical and/or radiological; RECIST 1.1 criteria) determined by the investigator, or date of death (whatever the cause), whichever occurs first. Patients alive without progression will be censored at the date of last news.
Patients' health according the questionnary quality of life C30 of EORTC | time between the date of the first dose treatment with tislelizumab and the date within the 30 days after the last dose of treatment
  Quality of life will be assessed with the questionnary quality of life C30 of EORTC (version 3.0) at each evaluation. Each questionnaire will be scored according to the relevant scoring manual. If half or more of the elements, which calculate a scale, are missing then the scale will be set to missing as per the scoring manuals. A scale cannot be estimated for the single item scales if the question they relate to has not been answered
Patients' health according the questionnary quality of life OES-18 of EORTC | time between the date of the first dose treatment with tislelizumab and the date within the 30 days after the last dose of treatment
  Quality of life will be assessed with the questionnary quality of life OES-18 of EORTC at each evaluation. Each questionnaire will be scored according to the relevant scoring manual. If half or more of the elements, which calculate a scale, are missing then the scale will be set to missing as per the scoring manuals. A scale cannot be estimated for the single item scales if the question they relate to has not been answered
Patients' health according the questionnary quality of life ELD14 of EORTC | time between the date of the first dose treatment with tislelizumab and the date within the 30 days after the last dose of treatment
  Quality of life will be assessed with the questionnary quality of life ELD14 of EORTC at each evaluation. Each questionnaire will be scored according to the relevant scoring manual. If half or more of the elements, which calculate a scale, are missing then the scale will be set to missing as per the scoring manuals. A scale cannot be estimated for the single item scales if the question they relate to has not been answered
Geriatric assessment according the questionnary G-CODE | time between the date of the first dose treatment with tislelizumab and the date within the 30 days after the last dose of treatment
  Geriatric assessment will be performed at baseline and during treatment using the complete G-CODE which assesses the patient's autonomy in their daily life
Prognostic value of immune biomarkers | the time between the date of the first dose treatment with tislelizumab and the first radiological tumoral evaluation at 9 weeks after C1J1
  All patients, participating in the clinical study, will have blood drawn for the biological assessments at baseline and at the first radiological tumoral evaluation.

CONTACTS AND LOCATIONS:
Locations (20):
- France (20):
  - Centre Hospitalier Annecy Genevois, Annecy, Epagny Metz-Tessy
  - Institut régional du cancer Provence d'Avignon, Avignon
  - Centre Hospitalier de la Côte Basque, Bayonne
  - CHU Besançon, Besançon
  - CH Béthune et Beuvry, Beuvry
  - ICHF Centre Pierre Curie, Beuvry
  - CHU Clermont-Ferrand, Clermont-Ferrand
  - CHU Dijon, Dijon
  - Groupe Hospitalier Mutualiste, Grenoble
  - CHRU Lille, Lille
  - CHU Limoges, Limoges
  - CHU Nancy, Nancy
  - Centre hospitalier de Perpignan, Perpignan
  - Centre Régional du Lutte Contre Le Cancer - Institut Godinot, Reims
  - CHU Rennes, Rennes
  - Institut de Cancérologie de l'Ouest, Saint-Herblain
  - Groupe Hospitalier Rance Emeraude, St-Malo
  - ICAN Strasbourg, Strasbourg
  - CHRU Tours, Tours
  - Médipôle Hôpital Mutualiste, Villeurbanne

IPD SHARING:
Plan to Share IPD: No